CLINICAL TRIAL: NCT05904405
Title: Perceived Quality of Family Planning Counseling and Its Determinants Among Reproductive Aged Women in El-dakhla District, New Valley Government,Egypt
Brief Title: Perceived Quality of Family Planning Counselling
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samah Ali Ezzat Mahmoud, Assistant Specialest at Obstetrics and Gynecology Department,Eldakhla General Hospital,New Valley Governorat. ., Assiut University
Other Study IDs: quality of family planning
Record Dates: First submitted 2023-03-28; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Contraception
Keywords: Counselling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: quationaire — Data will be collected through a semi-structured interview administered questionnaire which includes:
  1. Socio-demographic characteristics of women
  2. Family planning practice: This will include number of living children, current use of FP method and its type, and suggested causes of discontinuation of FP, previous contraceptive use, and reason for the visit 3-Facility factors such as gender of providers, qualification of providers, type of the health facility.
  4-Quality of contraceptive counseling (QCC) scale: it is a 22-item scale which measures the quality of care received by women during family planning visits. It includes : 1) information exchange, 2) interpersonal relations, and 3) disrespect and abuse in contraceptive counseling. The information exchange subscale consists of ten items, the interpersonal relationship subscale consists of seven items, and the disrespect and abuse subscale consists of five items.

SUMMARY:
The goal of this cross sectional study is to test Perceived quality of family planning counseling and its determinants among females in reproductive age in El-Dakhla District, New Valley government ,Egypt.

The main question[s] it aims to answer are:

1. During the contraception consultation, I was able to give my opinion about what I needed.
2. I received complete information about my options for contraceptive methods.
3. The provider knew how to explain contraception clearly.
4. I had the opportunity to participate in the selection of a method.
5. I received information about how to protect myself from sexually transmitted infections.
6. I received information about what to do if a method fails (e.g., broken condom, forget a pill, feel an IUD is poorly placed).
7. I could understand how my body might react to using contraception.
8. I could understand how to use the method(s) we talked about during the consultation.
9. I received information about what to do if I wanted to stop using a method.
10. The provider explained to me what to do if I had a reaction to a method (e.g., allergies, nausea, pains, menstrual changes).
11. I felt the information I shared with the provider was going to stay between us.
12. The provider gave me the time I needed to consider the contraceptive options we discussed.
13. The provider was friendly during the contraception consultation.
14. I felt the health care provider had sufficient knowledge about contraceptive methods.
15. The provider showed interest in my health while we talked about contraception.
16. The provider was interested in my opinions.
17. I felt listened to by the provider
18. The provider pressured me to use the method they wanted me to use.
19. I felt the provider treated me poorly because they tend to judge people.
20. I felt scolded because of my age.
21. The provider made me feel uncomfortable because of my sex life (e.g., when I started having sex, my sexual preferences, the number of partners I have, the number of children I have).
22. The provider looked at me or touched me in a way that made me feel uncomfortable.

DETAILED DESCRIPTION:
In 2017, Holt, Dehlendorf, and Langer created a framework for contraceptive counseling quality grounded in quality of care and human rights principles and research in healthcare communication.

Based on this framework, Holt et al. developed and validated the Quality of Contraceptive Counseling (QCC) Scale, which covers three interrelated aspects of counseling quality: information exchange, interpersonal relationship, and disrespect and abuse . The scale comprehensively measures aspects of the counseling process related not only to information receipt but also individuals' experiences having the opportunity to participate in the method selection process and the degree to which they had positive and trusting experiences with the provider .

Associations between quality of contraceptive counseling and characteristics of clients, such as age, education, and reproductive status, could represent significant health disparities and indicate the need for research. This study will seek to understand quality of family planning counseling utilizing the validated and client-centered based QCC Scale as experienced by reproductive aged women in El-Dakhla District, New Valley. Furthermore, it will investigate their associated factors either client, provider, or visit factors.

Data collection tool

Data will be collected through a semi-structured interview administered questionnaire which includes:

1. Socio-demographic characteristics of women such as age, education, occupation, religion, residence, husband's education, husband's occupation.
2. Family planning practice: This will include number of living children, current use of FP method and its type, and suggested causes of discontinuation of FP, previous contraceptive use, and reason for the visit

3-Facility factors such as gender of providers, qualification of providers, type of the health facility (mobile clinics???) 4-Quality of contraceptive counseling (QCC) scale: it is a 22-item scale which measures the quality of care received by women during family planning visits. It includes : 1) information exchange, 2) interpersonal relations, and 3) disrespect and abuse in contraceptive counseling. The information exchange subscale consists of ten items, the interpersonal relationship subscale consists of seven items, and the disrespect and abuse subscale consists of five items. Item responses were given on four-point Likert scales. Response categories for positively worded items were "completely agree" (4), "agree" (3), "disagree" (2), and "completely disagree" (1). Response categories for negatively worded items were "yes" (1), "yes with doubts" (2), "no with doubts" (3), and "no" (4). Composite subscale and total scores were calculated as mean scores .

Items of QCC scale:

Information exchange factor

1. During the contraception consultation, I was able to give my opinion about what I needed.
2. I received complete information about my options for contraceptive methods.
3. The provider knew how to explain contraception clearly.
4. I had the opportunity to participate in the selection of a method.
5. I received information about how to protect myself from sexually transmitted infections.
6. I received information about what to do if a method fails (e.g., broken condom, forget a pill, feel an IUD is poorly placed).
7. I could understand how my body might react to using contraception.
8. I could understand how to use the method(s) we talked about during the consultation.
9. I received information about what to do if I wanted to stop using a method.
10. The provider explained to me what to do if I had a reaction to a method (e.g., allergies, nausea, pains, menstrual changes).

    Interpersonal relationship factor
11. I felt the information I shared with the provider was going to stay between us.
12. The provider gave me the time I needed to consider the contraceptive options we discussed.
13. The provider was friendly during the contraception consultation.
14. I felt the health care provider had sufficient knowledge about contraceptive methods.
15. The provider showed interest in my health while we talked about contraception.
16. The provider was interested in my opinions.
17. I felt listened to by the provider

    Response Options:

    Completely agree - 4 Agree - 3 Disagree - 2 Completely disagree - 1 Disrespect and abuse factor
18. The provider pressured me to use the method they wanted me to use.
19. I felt the provider treated me poorly because they tend to judge people.
20. I felt scolded because of my age.
21. The provider made me feel uncomfortable because of my sex life (e.g., when I started having sex, my sexual preferences, the number of partners I have, the number of children I have).
22. The provider looked at me or touched me in a way that made me feel uncomfortable.

Response Options:

Yes - 1 Yes with doubts - 2 No with doubts - 3 No - 4

Scoring Procedures:

Scores from the individual items are used to calculate a composite score using a simple mean, with higher scores indicating higher reported quality of services

Statistical analysis Data entry and analysis will be carried out using SPSS version 24. Descriptive statistics will be done in the form of frequencies, mean and SD then analytic statistics will be done as chi square, independent sample test and correlations tests. Values will be considered significant when P values are equal to or less than 0.05.

Pilot study

Before starting to collect data, a pilot study will be carried out to fulfill the following purposes:

1. Testing the questionnaire form and detecting any modification required.
2. Estimation of the time needed to fill the questionnaire.
3. Detection of the difficulties that may arise and how to deal with them. Implications of the study Results of proposed study will be disseminated to stakeholders to help in planning paper interventions to improve quality of family planning services in El-Dakhla District, New Valley

Ethical Considerations

1. The research proposal will be reviewed and approved by the Ethical Committee of Assiut Faculty of Medicine.
2. Administrative permission will be obtained from Directorate of health affairs in New Valley Governrate.
3. Informed written consent will be obtained from subjects before being included in the study.
4. Privacy and confidentiality of the data will be assured.

ELIGIBILITY:
Inclusion Criteria:

-reproductive aged women (either adapter, continuer, and switcher) and seeking FB services (last counseling session)

Exclusion Criteria:

* Women who do not meet the above criteria will be excluded from the present study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: There are 18 primary health care centers and one general hospital in El-Dakhla District, New Valley. The target population will be selected from the general hospital and primary health centers of El-Dakhla District. The number of women chosen in each primary health center and the main hospital will be proportional to the number of women served by the facility until reaching the estimated sample size. The questionnaire will be distributed by the researcher herself to all women of the selected centers except those who refuse to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Quality of family planning counseling in family planning services, among reproductive aged women in El-Dakhla District, New Valley governorate . | one year
  Client reported quality of family planning counseling at family planning services and its determinants among 423 women at reproductive age in El-Dakhla District, New Valley. at different primary health centers of El-Dakhla District and El-Dakhla general hospital.
  By using questionnaire QCC Scale (quality of contraceptive counseling scale) .

REFERENCES:
- See also: 1. World Health Organization (WHO). WHO Definition of Family Planning-Public Health. 2020. p. Available at: https:// www.publichealth.com.ng/who. — https://www.publichealth.com.ng/who-definition-of-family-planning/